CLINICAL TRIAL: NCT05831059
Title: A Randomized, Controlled, Double-blind, Multicenter, Sympathetic Ganglion, High-voltage Pulsed Radiofrequency Ablation of Peripheral Neuralgia in Patients With Diabetic Foot
Brief Title: A Sympathetic Ganglion, High-voltage Pulsed Radiofrequency Ablation of Peripheral Neuralgia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ke Ma, Principal Investigator, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: XH-23-004
Record Dates: First submitted 2023-03-15; First posted 2023-04-26 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-04

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A group (Experimental): First receive pulse radio frequency treatment and then receive sham operation treatment
  Interventions: Radiation: Pulsed radio frequency therapy; Other: sham operation
- B group (Active Comparator): First receive sham operation treatment and then receive pulse radio frequency treatment
  Interventions: Radiation: Pulsed radio frequency therapy; Other: sham operation

INTERVENTIONS:
Radiation: Pulsed radio frequency therapy — Pulse Radio Frequency mode is a high voltage and low temperature Radio Frequency mode formed by discontinuous and pulsed current around nerve tissue
Other: sham operation — The means to achieve double-blind treatment had no practical effect on the subjects

SUMMARY:
The Sham Operation Group was used as control, the patients were assessed with the Digital Rating Scale (NRS) , the quality of life-related scale (Euro Qol) , clinical outcome measures: physician's overall impression of changes in pain (CGIC) and patient's overall impression change scale (PGIC) , skin temperature measurement, toe Oxygenation measurement, and anxiety and depression scores (Gad-7, Phq-9) , objective: to evaluate the efficacy and safety of high voltage pulsed radiofrequency in the treatment of peripheral neuralgia in patients with diabetic foot.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily participate in the study and sign the informed consent form;
* The age is between 18 (inclusive) and 85 (inclusive), regardless of gender;
* Body mass index (BMI) ≤ 45;
* Clinically diagnosed diabetes foot with moderate and severe pain in peripheral nerve of affected limb (defined as NRS score ≥ 4), the course of disease lasts for more than 12 months, and has been treated with clinical routine standard drugs (mecobalamin α- Lipoic acid, sodium valproate, carbamazepine, gabapentin/pregabalin, etc.) symptoms still exist at least 6 months later;
* Glycated hemoglobin<8%;
* Not participating in the drug/medical device test within 3 months before the test;

Exclusion Criteria:

* Patients who are in poor condition and cannot objectively describe symptoms or cooperate to complete the questionnaire score
* Ulcer is red and swollen, or active inflammatory infection;
* The affected limb has lesions such as blackening and gangrene of the toe skin;
* Those suffering from severe respiratory and cardiovascular diseases, liver and kidney insufficiency, and malignant tumors;
* Breast-feeding and pregnant women, or subjects with pregnancy plan within 1 month after the trial (also including male subjects);
* The daily dose of opioids is more than 120mg (different drug doses are converted into 120mg morphine sustained-release tablets);
* People with allergic diseases and allergic constitution;
* Have a history of drug abuse or drug addiction;
* There are contraindications to pulsed radio frequency therapy;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale | up to 4 months
  Numeric Rating Scale is the most widely used one-dimensional assessment scale，The higher the number, the more severe the pain

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai XINHUA Hospital, Shanghai, China